CLINICAL TRIAL: NCT04018521
Title: Use of Parent Connectors in First Episode Psychosis (FEP)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: inventional part of the study is registered under NCT05195489
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-00702; 18-A1-00-007376 (Other Grant/Funding Number: NATIONAL INSTITUTE OF MENTAL HEALTH (NIM))
Record Dates: First submitted 2019-07-09; First posted 2019-07-12 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: First Episode Psychosis (FEP)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent Connectors (Active Comparator): trained and supervised PPNs deliver weekly telephone-based support for six to nine months to parents or caregivers of all newlyenrolled youth or young adults (Y/YA) in FEP services
  Interventions: Behavioral: PPN; Behavioral: CSC Usual Care
- Usual Care (Active Comparator): Coordinated Specialty Care (CSC)
  Interventions: Behavioral: CSC Usual Care

INTERVENTIONS:
Behavioral: PPN — Delivery of Coordinated Specialty Care (CSC) for Y/YA in New York's state program for FEP, called OnTrackNY (OTNY).
  Arms: Parent Connectors
Behavioral: CSC Usual Care — standard of care provided to youth following first episode of psychosis

SUMMARY:
This study proposes to adapt an evidence based peer parent navigator (PPN) intervention, called Parent Connectors, in which trained and supervised PPNs deliver weekly telephone-based support for six to nine months to parents or caregivers of all newly enrolled youth or young adults (Y/YA) in FEP services. This PPN model will be used to enhance the delivery of Coordinated Specialty Care (CSC) for Y/YA in New York's state program for FEP, called OnTrackNY (OTNY). This research project has potential to add value to the CSC model through the inclusion of a feasible, low burden intervention that may improve family participation in services and Y/YA outcomes. Using random assignment, this study will examine the feasibility and preliminary impact of an accelerator strategy-the inclusion of peer parent navigators or PPNs-in CSC teams.

ELIGIBILITY:
Inclusion Criteria:

* Parents or caregivers of all newlyenrolled youth or young adults (Y/YA) in FEP services

Exclusion Criteria:

* NA

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Family Empowerment Scale (FES) | 9 Months
  A 34 item self reported instrument designed to measure empowerment status. The scale measures levels of empowerment, such as family, service system and community, and is rated on a likert scale, scale, ranging from1 (not true at all) to 5 (very true). The FES produces scores for three subscales based on level of empowerment:Family (12 items), Service system (12 items), and Community/ Political (10 items).
Patient Activation Measure (PAM) | 9 Months
  100-point quantifiable scale determining patient engagement in healthcare

IPD SHARING:
Plan to Share IPD: No